CLINICAL TRIAL: NCT03651622
Title: Accelerating Solutions to Optimize Glycemic Control and Weight Management In Young Adults With Type 1 Diabetes
Brief Title: ACT1ON Phase 2 (SMART Pilot) and Phase 3 (Efficacy Trial Development)
Acronym: ACT1ON DP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-1025; 1DP3DK113358-01 (NIH)
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 1; Overweight and Obesity
Keywords: Type 1 diabetes; T1D; Type 1 diabetes mellitus (T1DM); weight management; overweight; obese
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight; Obesity | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted; Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: This initial pilot and feasibility study uses a Sequential, Multiple Assignment, Randomized Trial (SMART) design to identify acceptable and effective dietary strategies to optimize both glycemic control and weight management. The study will be done at UNC and Stanford. Sequential randomization will occur at 0, 3.5, and 7 months. Following the baseline measurement visit and two week run-in period, participants will be randomized to one of three diets (stratified by site with block size of 4). Using a priori decision rules at 3.5 and 7 months post-initial randomization, those for whom the assigned diet is not acceptable or effective will be re-randomized (or re-assigned if only one diet remains untried). 10.5 months of follow-up time allows for evaluation of the effect of diets on initial weight loss and on early maintenance of initial weight loss. Decision criteria for re-randomization will incorporate clinical outcomes (glycemic control and weight change) and acceptability of the diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypocaloric, low carbohydrate (Experimental): Behavioral intervention to include lifestyle counseling on hypocaloric, low carbohydrate diet (15-20% calories from carbohydrate, 59-63% as total fat (<10% saturated fat, at least 37% monounsaturated fat, remaining as polyunsaturated fat). Using a priori decision rules at 3.5 and 7 months post-initial randomization, those for whom the diet assigned is not acceptable or is not effective will be re-randomized.
  Interventions: Behavioral: Hypocaloric, low carbohydrate diet
- Hypocaloric, moderate low fat (Experimental): Behavioral intervention to include lifestyle counseling on hypocaloric, moderate low fat diet (30% calories from fat) weight management based on the Look AHEAD study. Using a priori decision rules at 3.5 and 7 months post-initial randomization, those for whom the diet assigned is not acceptable or is not effective will be re-randomized.
  Interventions: Behavioral: Hypocaloric, moderate low fat diet
- Mediterranean, no caloric restriction (Experimental): Behavioral intervention to include lifestyle counseling on selecting a healthy Mediterranean diet, no caloric restriction. Using a priori decision rules at 3.5 and 7 months post-initial randomization, those for whom the diet assigned is not acceptable or is not effective will be re-randomized.
  Interventions: Behavioral: Mediterranean diet, no caloric restriction

INTERVENTIONS:
Behavioral: Hypocaloric, low carbohydrate diet — Participants will be advised on use of a hypocaloric, low carbohydrate diet using lifestyle counseling to include motivational interviewing and problem solving skills training strategies.
  Other Names: Low carbohydrate diet
  Arms: Hypocaloric, low carbohydrate
Behavioral: Hypocaloric, moderate low fat diet — Participants will be advised on use of a hypocaloric, moderate low fat diet using lifestyle counseling to include motivational interviewing and problem solving skills training strategies.
  Other Names: Low fat diet
  Arms: Hypocaloric, moderate low fat
Behavioral: Mediterranean diet, no caloric restriction — Participants will be advised on use of a healthy Mediterranean-based eating plan using lifestyle counseling to include motivational interviewing and problem solving skills training strategies.
  Other Names: Mediterranean diet
  Arms: Mediterranean, no caloric restriction

SUMMARY:
An initial pilot and feasibility study will be conducted using a Sequential, Multiple Assignment, Randomized Trial (SMART) design to identify acceptable and effective dietary strategies to optimize both glycemic control and weight management in young adults with Type 1 diabetes (T1D). This pilot trial will include a ten-and-a-half month behavioral intervention, with co-primary outcomes of glycemic control (HbA1C and hypoglycemia) and weight loss. The pilot trial will assess acceptability and adherence to three distinct, evidence-based dietary approaches designed to address weight management and glycemic control. Behavioral counseling strategies, use of carbohydrate counting for insulin dosing, and encouragement of physical activity will be the same across the three dietary approaches.

COVID-19 PROVISIONS: Due to restrictions in place on in-person visits due to COVID-19 precautions, some subjects may remain in the study longer than 10.5 months. As of June 2020, the study transitioned to a completely virtual format. Those who were due for a measurement visit during the time that research activities were halted, prior to the approval of the virtual procedures, remained on the diet they were currently assigned to, supported by bi-weekly Registered Dietitian (RD) counseling, until they were able to be scheduled for a virtual visit.

DETAILED DESCRIPTION:
Eight-four participants will be randomized in total; 42 at the University of North Carolina (UNC), 42 at Stanford.

COVID-19 Provisions: Due to impacts of COVID-19, the study was forced to cease recruitment early. 40 subjects were randomized at UNC and 29 were randomized at Stanford, for a total of 69 subjects across sites.

Procedures (methods):

Three distinct dietary approaches will be tested. Dietary approaches are as follows:

Diet 1: hypocaloric, moderate low fat (30% calories from fat) weight management based on the Look AHEAD study Diet 2: hypocaloric, low carbohydrate (15-20% calories from carbohydrate, 59-63% as total fat (<10% saturated fat, at least 37% monounsaturated fat, remaining as polyunsaturated fat) Diet 3: advice to select a healthy Mediterranean dietary pattern with no caloric restriction

Participants will complete measurement visits at baseline (-14 days), 3 mos, 6.5 mos, and 10 mos. All visits transitioned to a virtual format as of 6/2020 due to COVID-19 provisions.

Participants will complete a total of 23 intervention sessions over an approximately 10-and-a-half month period (Eight longer sessions (teleconference) and 15 telephone check-ins)

Participants will be randomized to one of the three diets for a minimum of a three-and-a-half month period. Re-randomization is possible following the 3 month and/or 6.5 month measurement visits. Re-randomization is based on acceptability of diet (self-report), non-severe hypoglycemic events (self-report), and not achieving significant weight change (defined as losing at least 2% of body weight from previous study visit), and worsening glycemic control (increase in Hemoglobin A1c of >/= 0.5% from previous study visit). Re-randomization will occur after the 14-day continuous glucose monitoring (CGM) wear period that will be initiated at each measurement visit.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 19-30 years old at enrollment
* History of Type 1 diabetes for greater than one year
* Latest hemoglobin A1c less than 13%
* BMI of 27-39

Exclusion Criteria:

* Individuals with other metabolic disorders, unstable thyroid disease, diagnosed eating disorder, prohibitive strict dietary restrictions or those with other serious condition that renders participation inappropriate
* Individuals who have experience diabetic ketoacidosis (DKA) or severe hypoglycemia requiring outside assistance in the last 6 months
* Females who are pregnant, breastfeeding, have delivered a baby in the last 12 months, or are planning to become pregnant during the study period.
* Individuals unwilling to follow any of the three study diets
* Individuals who monitor blood glucose less than 3 times a day

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mayer-Davis, PhD, Principal Investigator — UNC Chapel Hill; David M Maahs, MD, PhD, Principal Investigator — Stanford University; Richard Pratley, MD, Principal Investigator — Florida Hospital, Translational Research Institute
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Igudesman D, Crandell J, Corbin KD, Muntis F, Zaharieva DP, Casu A, Thomas JM, Bulik CM, Carroll IM, Pence BW, Pratley RE, Kosorok MR, Maahs DM, Mayer-Davis EJ. The Intestinal Microbiota and Short-Chain Fatty Acids in Association with Advanced Metrics of Glycemia and Adiposity Among Young Adults with Type 1 Diabetes and Overweight or Obesity. Curr Dev Nutr. 2022 Oct 30;6(10):nzac107. doi: 10.1093/cdn/nzac107. eCollection 2022 Nov. PMID 36349343
- [Derived] Muntis FR, Igudesman D, Sarteau AC, Thomas J, Arrizon-Ruiz N, Hooper J, Addala A, Crandell JL, Riddell MC, Maahs DM, Pratley RE, Corbin K, Mayer-Davis EJ, Zaharieva DP; ACT1ON Consortium. Relationship Between Moderate-to-Vigorous Physical Activity and Glycemia Among Young Adults with Type 1 Diabetes and Overweight or Obesity: Results from the Advancing Care for Type 1 Diabetes and Obesity Network (ACT1ON) Study. Diabetes Technol Ther. 2022 Dec;24(12):881-891. doi: 10.1089/dia.2022.0253. PMID 35984327
- [Derived] Corbin KD, Igudesman D, Addala A, Casu A, Crandell J, Kosorok MR, Maahs DM, Pokaprakarn T, Pratley RE, Souris KJ, Thomas JM, Zaharieva DP, Mayer-Davis EJ; ACT1ON Consortium. Design of the Advancing Care for Type 1 Diabetes and Obesity Network energy metabolism and sequential multiple assignment randomized trial nutrition pilot studies: An integrated approach to develop weight management solutions for individuals with type 1 diabetes. Contemp Clin Trials. 2022 Jun;117:106765. doi: 10.1016/j.cct.2022.106765. Epub 2022 Apr 20. PMID 35460915

RESULTS

PARTICIPANT FLOW:
Period: Diet Period 1 (Randomization 1)
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Started | 23 | 24 | 21
Completed | 19 | 17 | 12
Not Completed | 4 | 7 | 9
Not completed — Lost to Follow-up | 0 | 6 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 7
Period: Diet Period 2 (Randomization 2)
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Started | 19 | 15 | 14
Number of Participants Rerandomized From Hypocaloric, Low Carbohydrate Diet | 0 | 5 | 5
Number of Participants Rerandomized From Hypocaloric, Moderate Low Fat Diet | 5 | 0 | 6
Number of Participants Rerandomized From Mediterranean, no Caloric Restriction Diet | 5 | 4 | 0
Number of Participants Not Rerandomized | 9 | 6 | 3
Completed | 17 | 13 | 11
Not Completed | 2 | 2 | 3
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 0
Period: Diet Period 3 (Randomization 3)
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Started | 14 | 9 | 18
Number of Participants Rerandomized From Hypocaloric, Low Carbohydrate Diet | 0 | 2 | 10
Number of Participants Rerandomized From Hypocaloric, Moderate Low Fat Diet | 4 | 0 | 6
Number of Participants Rerandomized From Mediterranean | 6 | 4 | 0
Number of Participants Not Rerandomized | 4 | 3 | 2
Completed | 14 | 9 | 17
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction | Total
Number analyzed (Participants) | 23 | 24 | 21 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (3.3) | 24.9 (2.8) | 26.1 (3.2) | 25.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 20 | 49
  Male | 8 | 10 | 1 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 4 | 11
  Not Hispanic or Latino | 21 | 19 | 17 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 1 | 2 | 6
  White | 17 | 19 | 13 | 49
  More than one race | 1 | 1 | 4 | 6
  Unknown or Not Reported | 1 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 24 | 21 | 68
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 86.2 (10.7) | 91.9 (15.4) | 90.2 (15.6) | 89.4 (14.0)
Hemoglobin A1c (%) [Mean (Standard Deviation); unit: percent glycated hemoglobin] | 7.3 (1.5) | 8.2 (1.3) | 8.2 (1.3) | 7.9 (1.4)
Body fat [Median (Inter-Quartile Range); unit: Percent body fat] | 39.4 [27.1 to 45.1] | 39.8 [32.5 to 44.4] | 41.6 [36.9 to 45.2] | 40.4 [34.2 to 44.9]
Time in clinical hypoglycemia [Median (Inter-Quartile Range); unit: Percent of time] — 54-69 mg/dL Population: N's are smaller than the numbers initially randomized due to missing continuous glucose monitoring data.
  Percent of time
    number analyzed (Participants) | 19 | 22 | 17 | 58
    (all) | 3.5 [1.7 to 9.3] | 3.3 [1.4 to 5.5] | 4.1 [1.2 to 4.9] | 3.6 [1.6 to 5.6]
Time in target glucose range [Mean (Standard Deviation); unit: Percent of time] — 70-180 mg/dL Population: N's are smaller than the numbers initially randomized due to missing continuous glucose monitoring data.
  Percent of time
    number analyzed (Participants) | 19 | 22 | 17 | 58
    (all) | 54.1 (23.5) | 48.1 (19.3) | 48.0 (23.0) | 50.0 (21.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight - Randomization 1
Description: Weight in kilograms will be obtained at measurement visits at the beginning and end of this three-and-a-half month time period.
Time Frame: Baseline (-14 Days prior to Randomization 1 Visit), 3 Month (Measurement 2) Visit
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 19 | 17 | 12
kilograms | -1.6 (3.4) | -1.8 (5.7) | -1.5 (3.2)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.98, ANOVA

2. Primary Outcome: Change in Weight - Randomization 2
Description: as for outcome 1
Time Frame: 3 Month (Measurement 2) Visit, 6.5 Month (Measurement 3) Visit
Population: Completers for each diet period were participants who had sufficient data to be rerandomized. However, one participant on the Mediterranean diet who had insufficient data to be rerandomized had available weight data and was included in the weight analysis. Therefore, there is one more participant assigned to the Mediterranean diet for the weight analysis.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 17 | 13 | 12
kilograms | 0.27 (3.8) | 0.99 (4.1) | 0.86 (3.0)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.85, ANOVA

3. Primary Outcome: Change in Weight - Randomization 3
Description: as for outcome 1
Time Frame: 6.5 Month (Measurement 3) Visit, 10 Month (Measurement 4) Visit
Population: Data for one participant on the Mediterranean diet was excluded from analysis.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 14 | 9 | 16
kilograms | 0.68 (2.4) | -0.85 (2.3) | -0.64 (3.4)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.40, ANOVA

4. Primary Outcome: Change in HbA1C - Randomization 1
Description: HbA1c will be measured from a blood sample collected from participants. Blood will be obtained at measurement visits at the beginning and end of this three-and-a-half month time period.
Time Frame: Baseline (-14 Days prior to Randomization 1 Visit), 3 Month (Measurement 2) Visit
Measure: Mean (Standard Deviation); unit: Percent glycated hemoglobin
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 19 | 17 | 12
Percent glycated hemoglobin | -0.03 (0.55) | -0.48 (0.83) | 0.37 (0.88)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.02, ANOVA

5. Primary Outcome: Change in HbA1C - Randomization 2
Description: as for outcome 4
Time Frame: 3 Month (Measurement 2) Visit, 6.5 Month (Measurement 3) Visit
Measure: Mean (Standard Deviation); unit: Percent glycated hemoglobin
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 17 | 13 | 11
Percent glycated hemoglobin | -0.11 (0.65) | -0.008 (0.52) | -0.36 (0.66)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.38, ANOVA

6. Primary Outcome: Change in HbA1C - Randomization 3
Description: as for outcome 4
Time Frame: 6.5 Month (Measurement 3) Visit, 10 Month (Measurement 4) Visit
Measure: Mean (Standard Deviation); unit: Percent glycated hemoglobin
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 14 | 9 | 17
Percent glycated hemoglobin | 0.25 (0.72) | 0.72 (1.7) | -0.16 (0.74)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.18, ANOVA

7. Primary Outcome: Change in Time in Clinical Hypoglycemia - Randomization 1
Description: Change in the percent of time spent in clinical hypoglycemia (54-69 mg/dl) during Continuous Glucose Monitor (CGM) wear time will be assessed between the two weeks of wear from CGM insertion at Baseline Visit (-14 days) and the two weeks of wear from the insertion of the CGM at Measurement Visit 2.
Time Frame: 2 weeks of wear from Baseline Visit (-14 Days), 2 weeks of wear from 3 Month (Measurement 2) Visit
Population: The number of participants analyzed is fewer than the number of participants who completed the randomization period in each diet group due to missing data for continuous glucose monitoring.
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 15 | 13 | 9
Percent of time | -0.30 (4.1) | 0.65 (5.4) | -0.45 (1.7)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.79, ANOVA

8. Primary Outcome: Change in Time in Clinical Hypoglycemia - Randomization 2
Description: Change in the percent of time spent in clinical hypoglycemia (54-69 mg/dl) during CGM wear time will be assessed between the two weeks of wear from CGM insertion at Measurement 2 Visit and from CGM insertion at Measurement 3 Visit.
Time Frame: 2 weeks of wear from 3 Month (Measurement 2) Visit, 2 weeks of wear from 6.5 Month (Measurement 3) Visit
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 13 | 12 | 9
Percent of time | 0.2 (3.2) | 1.4 (4.2) | 2.6 (4.9)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; The proposed sample size of n=72 was sufficient to ensure 60% power to detect a moderate effect size (Cohen h=0.68) and 80% to detect a large effect size (Cohen h=0.85) at a significance level of 0.10 for comparing difference in change among the 3 diets. By design, our primary goal for this pilot work is to inform the final efficacy design of a fully powered SMART, and the pilot SMART was therefore not designed to be fully powered for all analyses; Test type: Superiority; p = 0.39, ANOVA

9. Primary Outcome: Change in Time in Clinical Hypoglycemia - Randomization 3
Description: Change in the percent of time spent in clinical hypoglycemia (54-69 mg/dl) during CGM wear time will be assessed between the two weeks of wear from CGM insertion at Measurement 3 Visit and from CGM insertion at Measurement 4 Visit.
Time Frame: 2 weeks of wear from 6.5 Month (Measurement 3) Visit, 2 weeks of wear from 10 Month (Measurement 4) Visit
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 13 | 8 | 15
Percent of time | 0.086 (2.5) | 0.97 (4.4) | -0.47 (5.3)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.75, ANOVA

10. Secondary Outcome: Change in Body Fat - Randomization 1
Description: Percent fat mass and percent fat free mass were measured via a dual-energy x-ray absorptiometry (DXA) scan at the beginning and end of this time three-and-a-half-month time period.
  COVID-19 PROVISIONS: Due to precautions required to prevent the spread of COVID-19, all in-person visits were discontinued as of 3/25/2020. As of this date, DXA scans at both sites were discontinued. Analysis on existing data continued, but no new DXA data were collected.
Time Frame: Baseline (-14 Days prior to Randomization 1 Visit), 3 Month (Measurement 2) Visit
Population: The number of participants analyzed is fewer than the number of participants who completed the randomization period in each diet group due to missing data for dual-energy x-ray absorptiometry, which was discontinued following the transition to a virtual protocol due to COVID-19.
Measure: Mean (Standard Deviation); unit: Percent body fat
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 16 | 12 | 10
Percent body fat | -0.87 (1.5) | -0.058 (1.2) | -0.57 (1.8)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.66, ANOVA

11. Secondary Outcome: Change in Body Fat - Randomization 2
Description: as for outcome 10
Time Frame: 3 Month (Measurement 2) Visit, 6.5 Month (Measurement 3) Visit
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of body fat
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 4 | 4 | 4
Percentage of body fat | -0.38 (2.7) | -0.28 (1.7) | 0.05 (2.1)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.96, ANOVA

12. Secondary Outcome: Change in Body Fat - Randomization 3
Description: as for outcome 10
Time Frame: 6.5 Month (Measurement 3) Visit, 10 Month (Measurement 4) Visit
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent body fat
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 2 | 1 | 1
Percent body fat | 1.4 (0.7) | 0.1 | -0.9
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.34, ANOVA

13. Secondary Outcome: Change in Time in Target Glucose Range - Randomization 1
Description: Change in percent of time spent in a pre-defined range of relative euglycemia (70-180 mg/dl, for a person with Type 1 diabetes) during CGM wear time, will be assessed between the two weeks of wear from CGM insertion at Baseline Visit (-14 days) and the two weeks of wear from CGM insertion at Measurement Visit 2.
Time Frame: 2 weeks of wear from 3 Month (Measurement 2) Visit, 2 weeks of wear from 6.5 Month (Measurement 3) Visit
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 15 | 13 | 9
Percent of time | 6.3 (19.1) | 3.8 (15.1) | -0.96 (13.1)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.58, ANOVA

14. Secondary Outcome: Change in Time in Target Glucose Range - Randomization 2
Description: Change in percent of time spent in a pre-defined range of relative euglycemia (70-180 mg/dl, for a person with Type 1 diabetes) during CGM wear time, will be assessed between the two weeks of wear from CGM insertion at Measurement 2 Visit and from CGM insertion at Measurement 3 Visit.
Time Frame: 2 weeks of wear from 3 Month (Measurement 2) Visit, 2 weeks of wear from 6.5 Month (Measurement 3) Visit
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 13 | 12 | 9
Percent of time | -0.60 (14.5) | 0.90 (14.4) | 1.0 (9.0)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.95, ANOVA

15. Secondary Outcome: Change in Time in Target Glucose Range - Randomization 3
Description: Change in percent of time spent in a pre-defined range of relative euglycemia (70-180 mg/dl, for a person with Type 1 diabetes) during CGM wear time, will be assessed between the two weeks of wear from CGM insertion at Measurement 3 Visit and from CGM insertion at Measurement 4 Visit.
Time Frame: 2 weeks of wear from 6.5 Month (Measurement 3) Visit, 2 weeks of wear from 10 Month (Measurement 4) Visit
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
Number analyzed (Participants) | 13 | 8 | 15
Percent of time | -2.1 (19.0) | -18.4 (27.0) | 1.1 (14.3)
Statistical Analysis 1: Comparison: Hypocaloric, Low Carbohydrate vs Hypocaloric, Moderate Low Fat vs Mediterranean, no Caloric Restriction; Test type: Superiority; p = 0.08, ANOVA

ADVERSE EVENTS:
Time Frame: 10.5 months per the study design, although participants who did not complete the study prior to the pandemic were monitored for a mean of 12.7 months due to study delays resulting from the COVID-19 pandemic.
Arm/Group | Hypocaloric, Low Carbohydrate | Hypocaloric, Moderate Low Fat | Mediterranean, no Caloric Restriction
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/39 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/39 | 0/48
Other Adverse Events (participants affected / at risk) | 5/43 | 1/39 | 8/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypocaloric, Low Carbohydrate (N=43) | Hypocaloric, Moderate Low Fat (N=39) | Mediterranean, no Caloric Restriction (N=48)
Diabetic ketoacidosis (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypocaloric, Low Carbohydrate (N=43) | Hypocaloric, Moderate Low Fat (N=39) | Mediterranean, no Caloric Restriction (N=48)
Seizure - diagnosed epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea and diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough and shortness of breath (General disorders) | 1 (1) | 0 (0) | 1 (2)
Hyperglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Suspected pregnancy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Jaw inflammation - wisdom tooth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT03651622/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03651622/SAP_001.pdf